CLINICAL TRIAL: NCT01956201
Title: Efficacy and Safety of Fenofibrate Added on to Atorvastatin Compared With Atorvastatin in Mixed Hypercholesterolemic Patient: Multi Center, Randomized, Double-blind, Parallel-group, Therapeutic Confirmatory Study.
Brief Title: Efficacy and Safety of Fenofibrate Added on to Atorvastatin Compared With Atorvastatin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 146MHL13011
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Atorvastatin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 20mg, Fenofibrate 160mg (Experimental): Atorvastatin 20mg, Fenofibrate 160mg: po, q.d.
  Interventions: Drug: Atorvastatin 20mg; Drug: Fenofibrate 160mg
- Atorvastatin 20mg, Placebo (Active Comparator): Atorvastatin 20mg, Placebo for Fenofibrate 160mg po, q.d.
  Interventions: Drug: Atorvastatin 20mg; Other: Placebo (Fenofibrate 160 mg)

INTERVENTIONS:
Drug: Atorvastatin 20mg — [Atorvastatin Run-in Period] Take Atorvastatin 20mg 1 tablet once a day (after breakfast) [Treatment Period] Take Atrovastatin 20mg/Fenofibrate 160mg or Atorvastiatin 20mg/Placebo of Finofibrate 160mg 2 tablet once a day (after breakfast) [Extension Period] Take Atrovastatin 20mg, Fenofibrate 160mg 2 tablet once a day (after breakfast)
  Other Names: Lipilou Tab.
Drug: Fenofibrate 160mg — Refer to Intervention Description of Atorvastatin 20mg
  Arms: Atorvastatin 20mg, Fenofibrate 160mg
Other: Placebo (Fenofibrate 160 mg) — Refer to Intervention Description of Atorvastatin 20mg
  Other Names: Placebo
  Arms: Atorvastatin 20mg, Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Atorvastatin and Fenofibrate compared with atorvastatin monotherapy in mixed hypercholesterolemic patients.

DETAILED DESCRIPTION:
Multi center, randomized, double-blind, parallel-group, therapeutic confirmatory study

Primary Outcome Measure:

The mean percent change of Non-HDL Cholesterol [Time Frame: from baseline at week 8]

Secondary Outcome Measures:

The achievement rate of LDL-C<100mg/dl, Non-HDL-C<130mg/dl [Time Frame: from baseline at week 8] The mean percent change of LDL-C, HDL-C, TG, TC, Apo-AI, Apo-B [Time Frame: from baseline at week 4, 8] The mean percent change of Non-LDL-C/HDL-C, TC/HDL-C, LDL-C/HDL-C, Apo-B/Apo-AI [Time Frame: from baseline at week 4, 8] The mean percent change of Fibrinogen, hs-CRP [Time Frame: from baseline at week 4, 8] Safety evaluation [Time Frame: Treatment period and Extension period]

ELIGIBILITY:
Inclusion Criteria:

* >19 years old
* High risk patient to Coronary Heart Disease (applied to 1 or more CHD risk factor listed below)

  1. Patient with Coronary Heart Disease
  2. Patient with carotid artery disease, peripheral blood vessel disease, abdominal aneurysm
  3. Patient with diabetes(HbA1C≤9.0%)
  4. 10-year risk of CHD >20%(by Framingham 10-year risk score calculation)
* At Visit 1(Screening)

  1. 100mg/dl≥LDL-C, 150mg/dl≤TG≤500mg/dl

     * 4weeks of Atorvastatin 20mg monotherapy run-in period
  2. LDL-C<100mg/dl, 150mg/dl≤TG≤500mg/dl

     * If treated with Atorvastatin 20mg monotherapy 4weeks prior to this study
* At Visit 2(After 4weeks of Atorvastatin monotherapy run-in period)

  * LDL<100mg/dl, 150mg/dl≤TG≤500mg/dl

Exclusion Criteria:

* Patients with acute artery disease within 3 months
* Patients with congestive heart failure(NYHA class III~IV) or uncontrolled arrhythmia within 6 months
* Patients with uncontrolled hypertension(SBP>160mmHg or DBP>95mmHg)
* TSH>1.5X ULN
* Patients with myopathy, rhabdomyolysis or CK>2X ULN
* Hypersensitive to Atorvastatin and/or Fenofibrate or had photoallergy or phototoxicity during fibrate and/or ketoprofen treatment
* Serum Creatinine>2.5mg/dl, AST or ALT > 2X ULN
* History of drug or alcohol abuse within 6 months
* History of GI tract surgery or disability to drug absorption
* Women with pregnant, breast-feeding
* Patients with gallbladder disease
* Patients with biliary cirrhosis
* Patients with pancreatitis(acute pancreatitis is excluded due to severe hypertriglyceridemia)
* Patients treated with any investigational drugs within 4 weeks at the time consents are obtained
* History of malignant tumor including leukemia, lymphoma within 5 years
* Patients must be treated with medications prohibited for concomitant use during study period
* Not eligible to participate for the study at the discretion of investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The mean percent change of Non-HDL Cholesterol | from baseline at week 8

SECONDARY OUTCOMES:
The achievement rate of LDL-C<100mg/dl, Non-HDL-C<130mg/dl | from baseline at week 8
The mean percent change of LDL-C, HDL-C, TG, TC, Apo-AI, Apo-B | from baseline at week 4, 8
The mean percent change of Non-LDL-C/HDL-C, TC/HDL-C, LDL-C/HDL-C, Apo-B/Apo-AI | from baseline at week 4, 8
The mean percent change of Fibrinogen, hs-CRP | from baseline at week 4, 8
Safety evaluation (Physical examination, Vital sign, Laboratory, AE etc.) | Treatment period (8 weeks) and Extension period (16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: MoonKyu Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center - Seoul
Locations (30):
- South Korea (30):
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kangwon University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Dongguk University Ilsan Hospital, Ilsan
  - Inje University Ilsan Paik Hospital, Ilsan
  - Chonbuk National University Hospital, Jeonju
  - Hanyang University Guri Hospital, Kyunggi
  - Seoul National University Hospital, Bundang, Seongnam
  - Asan Medical Center, Seoul
  - Eulji General Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Huro Hospital, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Kyunghee University Medical center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Seoul
  - The Catholic University of korea, Yeouido St. Mary's Hospital, Seoul
  - Ajou University hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju